CLINICAL TRIAL: NCT01960764
Title: Phase 1 Study of Whether Host Preconditioning Modifies Short-term Transplant Survival
Brief Title: Examination of Whether Host Preconditioning Modifies Short-term Transplant Survival
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This sub-study was not done because main study results reached significance.
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Richard Gallo, Professor and Chief, Division of Dermatology, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSD 131244.2
Record Dates: First submitted 2013-09-30; First posted 2013-10-11 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Autologous microbiome transplant; Bacteria transplant; Treatment for atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-Treatment (Experimental): Prior to receiving the transplant, this arm will be washed with an antimicrobial regimen
  Interventions: Drug: Pre-Treatment with Dial liquid antibacterial soap
- Control (Placebo Comparator): This arm will still be transplanted with the autologous microbiome transplant cream, however it will not be pre-treated with an antimicrobial regimen
  Interventions: Other: Control

INTERVENTIONS:
Drug: Pre-Treatment with Dial liquid antibacterial soap — This arm will be pre-treated with Dial liquid antibacterial soap and alcohol prior to the autologous microbiome transplant.
  Arms: Pre-Treatment
Other: Control
  Other Names: This arm will not be pre-treated, but rather will have the autologous microbiome transplant cream applied without any pre-treatment regimen.
  Arms: Control

SUMMARY:
Unlike healthy control skin, the skin of patients with atopic dermatitis (AD) is frequently colonized by Staphylococcus aureus (S. aureus), putting these patients at increased risk of S. aureus skin infections. In addition, research in the investigator's lab has shown that these patients have fewer protective antimicrobial Staphylococcal species such as Staphylococcal epidermidis (S. epidermidis) known to produce antimicrobial peptides that play a role in protecting the skin from invading pathogens. In this study, the investigator will attempt to decrease S. aureus colonization and increase colonization by protective Staph species. First the investigator will culture the bacteria on subjects' lesional AD skin. The investigator will selectively grow the subject's antimicrobial Staph colonies and place them into a base moisturizer. The moisturizer plus bacteria will be applied to both of the subject's arms. Prior to applying this, though, one arm will first be pre-treated with an antimicrobial regiment of Dial liquid antibacterial soap and alcohol. We will then compare the abundance of antimicrobial Staph species on each subject's arms 24 hours later to determine whether the pre-treatment regimen increased survival of the transplanted antimicrobial Staph species. The investigator expects that the arm pre-treated with the antimicrobial regimen will have more antimicrobial Staph species at this time point.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects who are not pregnant or lactating
* 18-80 years of age
* Diagnosis of atopic dermatitis for at least 6 months using the Hanifin and Rajka Diagnostic Criteria for atopic dermatitis
* Presence of lesional atopic dermatitis skin in both antecubital fossae
* Positive S. aureus colonization based on results of a skin culture taken from one of their AD-affected antecubital fossae during the screening visit

Exclusion Criteria:

* Use of any topical AD treatments (including topical steroids, topical calcineurin inhibitors) to either arm within one week of either screening visit
* Use of any oral/systemic AD therapies (antihistamines, steroids) within 28 days of either screening visit
* Severe AD that would worsen significantly from holding a participant's usual topical/oral AD medications for the time periods required in the inclusion/exclusion criteria (one week prior to the screening visits and during the study for topical medications and 28 days prior to screening visits and during the study for oral medications)
* Subjects who have taken a bleach bath within a week prior to screening, or who take bleach baths during the study
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Subjects with Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
* Any subject who is immunocompromised (e.g. provides researchers with a history lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome) or has a history of malignant disease (with the exception of non-melanomatous skin cancer). This information will be gathered verbally from the patient while taking a medical history from the patient, and will not involve further testing such as an HIV test.
* Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
* Active bacterial, viral or fungal skin infections
* Any noticeable breaks or cracks in the skin on either arm, including severely excoriated skin or skin with open or weeping wounds suggestive of an active infection or increased susceptibility to infection.
* Ongoing participation in another investigational trial
* Use of any oral or topical antibiotic for up to four weeks prior to screening
* Use of any systemic immunosuppressive therapy (e.g. cyclosporine, methotrexate, etc.) within four weeks of screening.
* Sensitivity to or difficulty tolerating Dove fragrance-free bar soap, Dial antibacterial liquid soap, Cetaphil lotion, or alcohol-based cleaners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Abundance of antimicrobial Staph colonies | 24-hours post-transplant
  Quantitative washes will be used to measure the abundance of antimicrobial Staph colonies on both the pre-treated and the not pre-treated arms 24 hours after the microbial transplant

SECONDARY OUTCOMES:
Adverse events | 24 hours post-transplant
  All adverse events associated with use of the transplant cream will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States